CLINICAL TRIAL: NCT02725281
Title: Comparison of Two Different Distraction Methods Affecting the Level of Pain and Anxiety During Extracorporeal Shock Wave Lithotripsy
Brief Title: Pain and Anxiety During Extracorporeal Shock Wave Lithotripsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Elif Gezginci, RN, Msc, PhDs, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 50687469-1491-85-14/1648.4-464
Record Dates: First submitted 2016-03-14; First posted 2016-03-31 (Estimated); Last update posted 2024-12-03 (Actual); Status verified 2024-12

CONDITIONS: Urinary Tract Stones; Pain; Anxiety
MeSH Terms: conditions — Urinary Calculi; Pain; Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control group (No Intervention): The patients in "Group 1" didn't receive any intervention during ESWL.
- Stress ball (Active Comparator): The patients in "Group 2" were given stress ball into both their palms 5 minutes before ESWL. Participants were instructed to "squeeze the balls twice after counting up to ten" and "repeat it until the end of the procedure". This ball was medium hard and it was made of high quality silicon.
  Interventions: Other: Stress ball
- Music (Active Comparator): The patients in "Group 3" were listened to the music chosen by them with a headset as a nonpharmacological method during lithotripsy.
  Interventions: Other: Music

INTERVENTIONS:
Other: Stress ball — The patients in this group were given stress ball into both their palms 5 minutes before ESWL. Participants were instructed to "squeeze the balls twice after counting up to ten" and "repeat it until the end of the procedure". This ball was medium hard and has been made of high quality silicon.
  Arms: Stress ball
Other: Music — The patients in this group were also listened to the music chosen by them with a headset from 5 min before until the end of lithotripsy. Types of music played for the patients were Turkish folk music, Turkish art music, Turkish arabesque music, Turkish pop music, foreign pop music, rock music, and classical music.
  Arms: Music

SUMMARY:
Investigators observed that during the Extracorporeal Shock Wave Lithotripsy (ESWL) non-pharmacological methods used for reducing the level of the pain and anxiety among the patients with the urinary stones are not sufficient and the effectiveness of these methods is controversial. There are very few studies, which investigated the effects of music on the pain and anxiety during ESWL. In addition, any randomized clinical trial related to the use of stress ball for relaxation and distraction on the reduction of pain and anxiety during lithotripsy has not been found in the relevant literature. Investigators also evaluated that further evidence-based studies are necessary. Thus, investigators aimed to investigate the effectiveness of stress ball and music for reducing the pain and anxiety of the patients during ESWL in this study.

DETAILED DESCRIPTION:
Extracorporeal Shock Wave Lithotripsy (ESWL), used commonly in urinary stone treatment, can cause pain and anxiety for patients. The aim of this study was to investigate the efficacy of use of music and stress ball to reduce pain and anxiety during lithotripsy. This was a single center parallel-randomized controlled trial. The study sample consisted of a total of 120 patients who applied to lithotripsy unit of urology clinic in a training and research hospital in Turkey between April and September 2014. The patients were randomly divided into three groups. The patients in group-I (control group) were not interfered, while group-II was given stress ball into their palms in order to squeeze and group-III was listened to the music chosen by themselves with a headset during the lithotripsy procedure. Data were collected using the Patient Information Form, Visual Analogue Scale (VAS), and State Trait Anxiety Inventory (STAI-SA).

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria of this study were to have kidney or ureter stones eligible for the ESWL procedure based on the European Association of Urology Guideline,
* To be the first lithotripsy treatment,
* To be older than 18 years old,
* To have the body mass index of 30kg/m2 or less,
* Not to be given analgesic before the procedure,
* Not to have renal colic just before ESWL,
* Not to have any contraindication in terms of lithotripsy,
* Not to have ureteral stent.

Exclusion Criteria:

* To refuse to participate in this study,
* Not to meet the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
A change on pain severity in VAS (Visual Analogue Scale) pain scale reported by the patients at the end of lithotripsy procedure compared with the baseline | 5 min before and 5 min after the ESWL process
  Pain

SECONDARY OUTCOMES:
A change on anxiety level in STAI-SA (State-Trait Anxiety Inventory-State Anxiety) at the end of procedure compared with the baseline | 5 min before and 5 min after the ESWL process
  Anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Elif Gezginci, RN,PhDs, Principal Investigator — Saglik Bilimleri Universitesi Gulhane Tip Fakultesi; Emine Iyigun, RN,AssocProf, Study Director — Saglik Bilimleri Universitesi Gulhane Tip Fakultesi; Serdar Yalcin, MD, Principal Investigator — Saglik Bilimleri Universitesi Gulhane Tip Fakultesi; Selahattin Bedir, MD,Prof, Study Director — Saglik Bilimleri Universitesi Gulhane Tip Fakultesi; Yasar I. Ozgok, MD,Prof, Study Director — Saglik Bilimleri Universitesi Gulhane Tip Fakultesi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aboumarzouk OM, Kata SG, Keeley FX, McClinton S, Nabi G. Extracorporeal shock wave lithotripsy (ESWL) versus ureteroscopic management for ureteric calculi. Cochrane Database Syst Rev. 2012 May 16;2012(5):CD006029. doi: 10.1002/14651858.CD006029.pub4. PMID 22592707
- [Background] Akin Y, Yucel S. Long-term effects of pediatric extracorporeal shockwave lithotripsy on renal function. Res Rep Urol. 2014 Apr 28;6:21-5. doi: 10.2147/RRU.S40965. eCollection 2014. PMID 24892029
- [Background] Bosio, A., Destefanis, P., Buffardi, A., Alessandria, E., Dalmasso, E., Lucci Chiarissi, M., Berta, G., Bisconti, A., Fontana, D., & Frea, B. E68 Does music reduce discomfort during ESWL? A prospective randomized trial. European Urology Supplements, 2013 3;12:53.
- [Background] Cepeda MS, Diaz JE, Hernandez V, Daza E, Carr DB. Music does not reduce alfentanil requirement during patient-controlled analgesia (PCA) use in extracorporeal shock wave lithotripsy for renal stones. J Pain Symptom Manage. 1998 Dec;16(6):382-7. doi: 10.1016/s0885-3924(98)00099-2. PMID 9879163
- [Background] Coll AM, Ameen JR, Mead D. Postoperative pain assessment tools in day surgery: literature review. J Adv Nurs. 2004 Apr;46(2):124-33. doi: 10.1111/j.1365-2648.2003.02972.x. PMID 15056325
- [Background] Demir, Y. (2012). Non-pharmacological therapies in pain management. INTECH Open Access Publisher.
- [Background] Diana, K.J., & George, K.V. (2013). Urinary stone formation: Efficacy of seed extract of Ensete superbum (Roxb.) Cheesman on growth inhibition of calcium hydrogen phosphate dihydrate crystals. Journal of Crystal Growth, 363, 164-170.
- [Background] Joshi HN, Karmacharya RM, Shrestha R, Shrestha B, de Jong IJ, Shrestha RK. Outcomes of extra corporeal shock wave lithotripsy in renal and ureteral calculi. Kathmandu Univ Med J (KUMJ). 2014 Jan-Mar;12(45):51-4. doi: 10.3126/kumj.v12i1.13639. PMID 25219995
- [Background] Karabulut, N., Gürçayır, D., & Aktaş, Y.Y. (2015). Non-pharmacological interventions for pain management used by nursing students in Turkey. Kontakt.
- [Background] Lee DW, Chan KW, Poon CM, Ko CW, Chan KH, Sin KS, Sze TS, Chan AC. Relaxation music decreases the dose of patient-controlled sedation during colonoscopy: a prospective randomized controlled trial. Gastrointest Endosc. 2002 Jan;55(1):33-6. doi: 10.1067/mge.2002.120387. PMID 11756911
- [Background] Ngee-Ming G, Tamsin D, Rai BP, Somani BK. Complementary approaches to decreasing discomfort during shockwave lithotripsy (SWL). Urolithiasis. 2014 Jun;42(3):189-93. doi: 10.1007/s00240-014-0655-2. Epub 2014 Mar 20. PMID 24648110
- [Background] Öner, N., & Le Compte, A. (1985). Durumluk/Sürekli Kaygi Envanteri El Kitabı. (State-Trait Anxiety Inventory Handbook) 2. Baskı, Boğaziçi Üniversitesi Yayınları, Istanbul No:333, 52-56.
- [Background] Ozsaker E, Diramali A. The effect of transcutaneous electrical nerve stimulation for pain relief during extracorporeal shock-wave lithotripsy procedure. Pain Manag Nurs. 2014 Mar;15(1):59-68. doi: 10.1016/j.pmn.2012.06.003. Epub 2012 Aug 18. PMID 24602425
- [Background] Pearle, M.S., & Lotan, Y. (2012). Urinary lithiasis: etiology, epidemiology, and pathogenesis. Camphel-walsh Urology, 10, 1257-1286.
- [Background] Perera, N.D., & Perera S.J. (2013). The role of extracorporeal shock wave lithotripsy in renal calculi. Sri Lanka Journal of Surgery, 31(3), 33-40.
- [Background] Resim S, Gumusalan Y, Ekerbicer HC, Sahin MA, Sahinkanat T. Effectiveness of electro-acupuncture compared to sedo-analgesics in relieving pain during shockwave lithotripsy. Urol Res. 2005 Aug;33(4):285-90. doi: 10.1007/s00240-005-0473-7. Epub 2005 Jun 22. PMID 15971087
- [Background] Salinas AS, Lorenzo-Romero J, Segura M, Calero MR, Hernandez-Millan I, Martinez-Martin M, Virseda JA. Factors determining analgesic and sedative drug requirements during extracorporeal shock wave lithotripsy. Urol Int. 1999;63(2):92-101. doi: 10.1159/000030425. PMID 10592496
- [Background] Schade GR, Faerber GJ. Urinary tract stones. Prim Care. 2010 Sep;37(3):565-81, ix. doi: 10.1016/j.pop.2010.05.003. PMID 20705199
- [Background] Stevensen C. Non-pharmacological aspects of acute pain management. Complement Ther Nurs Midwifery. 1995 Jun;1(3):77-84. doi: 10.1016/s1353-6117(05)80081-2. PMID 9456714
- [Background] Turk, C., Knoll, T., Petrik, A., Sarica, K., Skolarikos, A., Straub, M., & Seitz, C. (2014). Guidelines on urolithiasis. European Association of Urology.
- [Background] Wang SM, Punjala M, Weiss D, Anderson K, Kain ZN. Acupuncture as an adjunct for sedation during lithotripsy. J Altern Complement Med. 2007 Mar;13(2):241-6. doi: 10.1089/acm.2006.6262. PMID 17388767
- [Background] Williamson A, Hoggart B. Pain: a review of three commonly used pain rating scales. J Clin Nurs. 2005 Aug;14(7):798-804. doi: 10.1111/j.1365-2702.2005.01121.x. PMID 16000093
- [Background] Yilmaz E, Ozcan S, Basar M, Basar H, Batislam E, Ferhat M. Music decreases anxiety and provides sedation in extracorporeal shock wave lithotripsy. Urology. 2003 Feb;61(2):282-6. doi: 10.1016/s0090-4295(02)02375-0. PMID 12597931